CLINICAL TRIAL: NCT07051616
Title: The Impact of Children Laughter Intervention on Anxiety, Nausea, Vomiting, and Fatigue in Chemotherapy Patients - A Randomized Controlled Trial
Brief Title: The Effect of Children's Laughter Video on Oncology Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sibel Küçükoğlu, Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/25
Record Dates: First submitted 2025-06-25; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Chemotherapy Effect; Laughter; Fatigue; Nausea; Vomiting
MeSH Terms: conditions — Anxiety Disorders; Laughter; Fatigue; Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child laughter video group (Experimental): Patients in this group were made to watch the laughter video prepared by the researchers at the end of the 1st and 2nd hour after the start of chemotherapy.
  Interventions: Behavioral: Child laughter video
- Control Group (No Intervention): Participants in the control group were not subjected to any intervention other than routine practice during chemotherapy.

INTERVENTIONS:
Behavioral: Child laughter video — 1 hour after the chemotherapy treatment was started, the video monitor was placed at a height where the patient could see comfortably while lying down and the video, which was checked and prepared beforehand, was turned on full screen. The appropriate volume was adjusted and the patient was allowed to watch the video for 10 minutes without any other intervention. The video was then stopped and the etagere was removed from in front of the patient. Chemotherapy was continued. At the 2nd hour of chemotherapy, the disinfected etagere and computer were placed in a position where the patient could see them comfortably and the 2nd video was started and the patient was allowed to watch the video for 10 minutes.
  Arms: Child laughter video group

SUMMARY:
This study was conducted to investigate the effect of video playback of children's laughter on anxiety, nausea, vomiting and fatigue levels of patients during chemotherapy

DETAILED DESCRIPTION:
Nausea and vomiting, anxiety and fatigue due to chemotherapy can be prevented or reduced with effective nursing interventions and care. Laughter therapy is an intervention that has been used in the symptom management of individuals with cancer in recent years. Studies focusing on humor and laughter have generally been conducted among cancer patients. Humor and laughter have been shown to have both physiological, psychological and sociological benefits for patients in general. When the studies on laughter yoga are examined, it is seen that the results of laughter therapy applied to individuals are examined. It has also been reported in the literature that laughter has a contagious effect, often occurring in groups of people. There is no study in the literature on the effect of children's laughter on adults. This study will reveal the effectiveness of infant and child laughter in patients receiving chemotherapy. It is thought that this study will constitute an important data source for experimental studies to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with lymphoma (preferred to have the same type of cancer)
* Receiving the R - Chop cycle protocol as chemotherapy (This cycle was preferred because of the nausea and vomiting experienced in this protocol and the duration of the treatment is 4-5 hours) (Cleveland Clinic 2025).
* Inpatient hospitalization,
* Be over 18 years of age,
* Conscious, oriented and cooperative

Exclusion Criteria:

* Don't take a different cure than R - Chop,
* Visual and hearing and cognitive impairment,
* Do not have a problem that creates a communication barrier,
* Having any psychiatric illness such as depression, euphoria and taking psychiatric medication
* Refusal to participate in the study
* Other non-pharmacological methods

Ages: 32 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Patient information form | First measurement-10. minutes before the start of the patient's chemotherapy
  The form was designed by the researchers in two parts to assess personal characteristics and characteristics related to the disease and treatment.
Spielberger State Anxiety Scale | First measurement- 5 minutes before the start of the patient's chemotherapy
  The scale measures the level of status anxiety of the patient with 20 questions.this form was applied in the pre-test and post-test phase
FACIT Fatigue Scale | First measurement- 1 minutes before the start of the patient's chemotherapy
  Developed by Singh in 2014, the scale was developed to evaluate the relationship between anemia and fatigue in cancer patients and to meet the increasing demand. This form was applied in the pre-test and post-test phase.
Physiological Parameter Follow-up Form (Heart rate-min) | As soon as chemotherapy is started (Within first five minute)
  This form was created by researchers. When chemotherapy started and measured at the beginning of each hour.
Physiological Parameter Follow-up Form (Respiration rate- min) | As soon as chemotherapy is started (Within first five minute)
  This form was created by researchers. When chemotherapy started and measured at the beginning of each hour.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | As soon as chemotherapy is started (Within first five minute)
  This form was created by researchers. When chemotherapy started and measured at the beginning of each hour.
Physiological Parameter Follow-up Form (blood pressure- mmHg) | As soon as chemotherapy is started (Within first five minute)
  This form was created by researchers. When chemotherapy started and measured at the beginning of each hour.
Nausea Follow-up Form | As soon as chemotherapy is started (Within first five minute)
  With this form, the presence or absence of the patient's nause was questioned.Nausea was first measured at the start of chemotherapy
Vomiting Follow-up Form | As soon as chemotherapy is started (Within first five minute)
  With this form, the presence or absence of the patient's vomiting was questioned. Vomiting was first measured at the start of chemotherapy

SECONDARY OUTCOMES:
Physiological Parameter Follow-up Form (Heart rate-min) | Second measurement: 1. hour after starting chemotherapy
  The measurement was made immediately after the first hour was full.
Physiological Parameter Follow-up Form (Respiration rate- min) | Second measurement: 1. hour after starting chemotherapy
  The measurement was made immediately after the first hour was full.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Second measurement: 1. hour after starting chemotherapy
  The measurement was made immediately after the first hour was full.
Physiological Parameter Follow-up Form (blood pressure- mmHg) | Second measurement: 1. hour after starting chemotherapy
  The measurement was made immediately after the first hour was full.
Nausea Follow-up Form | Second measurement: 1. hour after starting chemotherapy
  The measurement was made immediately after the first hour was full.
Vomiting Follow-up Form | Second measurement: 1. hour after starting chemotherapy
  The measurement was made immediately after the first hour was full.
Physiological Parameter Follow-up Form (Heart rate-min) | Third measurement: 2. hour after starting chemotherapy
  The measurement was made immediately after the second hour was full.
Physiological Parameter Follow-up Form (Respiration rate- min) | Third measurement: 2. hour after starting chemotherapy
  The measurement was made immediately after the second hour was full.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Third measurement: 2. hour after starting chemotherapy
  The measurement was made immediately after the second hour was full.
Physiological Parameter Follow-up Form (blood pressure- mmHg) | Third measurement: 2. hour after starting chemotherapy
  The measurement was made immediately after the second hour was full.
Nausea Follow-up Form | Third measurement: 2. hour after starting chemotherapy
  The measurement was made immediately after the second hour was full.
Vomiting Follow-up Form | Third measurement: 2. hour after starting chemotherapy
  The measurement was made immediately after the second hour was full.
Physiological Parameter Follow-up Form (Heart rate-min) | Fourth measurement: 3. hour after starting chemotherapy
  The measurement was made immediately after the third hour was full.
Physiological Parameter Follow-up Form (Respiration rate- min) | Fourth measurement: 3. hour after starting chemotherapy
  The measurement was made immediately after the third hour was full.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Fourth measurement: 3. hour after starting chemotherapy
  The measurement was made immediately after the third hour was full.
Physiological Parameter Follow-up Form (blood pressure- mmHg) | Fourth measurement: 3. hour after starting chemotherapy
  The measurement was made immediately after the third hour was full.
Nausea Follow-up Form | Fourth measurement: 3. hour after starting chemotherapy
  The measurement was made immediately after the third hour was full.
Vomiting Follow-up Form | Fourth measurement: 3. hour after starting chemotherapy
  The measurement was made immediately after the third hour was full.
Physiological Parameter Follow-up Form (Heart rate-min) | Fifth measurement: 4. hour after starting chemotherapy
  The measurement was made immediately after the fourth hour was full.
Physiological Parameter Follow-up Form (Respiration rate- min) | Fifth measurement: 4. hour after starting chemotherapy
  The measurement was made immediately after the fourth hour was full.
Physiological Parameter Follow-up Form (oxygen saturation -SpO2%) | Fifth measurement: 4. hour after starting chemotherapy
  The measurement was made immediately after the fourth hour was full.
Physiological Parameter Follow-up Form (blood pressure- mmHg) | Fifth measurement: 4. hour after starting chemotherapy
  The measurement was made immediately after the fourth hour was full.
Nausea Follow-up Form | Fifth measurement: 4. hour after starting chemotherapy
  The measurement was made immediately after the fourth hour was full.
Vomiting Follow-up Form | Fifth measurement: 4. hour after starting chemotherapy
  The measurement was made immediately after the fourth hour was full.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Prof, Principal Investigator — Selcuk University
Locations (1):
- Sibel Küçükoğlu, Selçuklu, Akademi Mahallesi, Turkey (Türkiye)